CLINICAL TRIAL: NCT00782743
Title: Prospective Comparison of Phenprocoumon (Marcumar) and Acetylsalicylic Acid (ASA)With Regard to the Progress of Valvular and Coronary Calcification
Brief Title: Comparison of Phenprocoumon and Acetylsalicylic Acid (ASA)
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Marcumar-ASS-Study; Eudra-CT-Number 2007-001685-33; Study-Number 07/002
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Valvular Calcification; Coronary Calcification
Keywords: phenprocoumon; anticoagulation; acetylic salicylic acid; Need for new anticoagulation treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers for inflammation, measuring of inhibitors of calcification
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with required new anticoagulation with phenprocoumon 1/2 of them with a GFR< 60 ml/min and >15 ml/min
- 2: patients with required therapy with ASS, 1/2 of them with a GFR <60 ml/min and >15 ml/min

SUMMARY:
In this open, prospective, non-randomised, parallel group, unicentric pilot-study will be compared the progress of valvular and coronary calcification with regard to the therapy with either acetyl-salicylic acid or phenprocoumon. The progress of calcification is documented by comparison of cardial stratified computed tomography. It is supposed that treatment with phenprocumon leads to increased coronary and valvular calcification as well to decreased blood levels of carboxylated matrix-GLA-protein

DETAILED DESCRIPTION:
Patients will be allocated to two groups with either

1. anticoagulation with phenprocoumon (needed for at least 1 year)
2. therapy with ASA

Both treatment groups should include to 50% patients with a glomerular filtration rate (GFR) < 60 ml/min and > 15 ml/min.

All patients will undergo a screening procedure with evaluation of calcium regulating proteins, echocardiography and stratified computed tomography of the heart. Medical check up's are planned after 1,3,6, 12 and 18 months.

Prior investigations concern diastolic ventricular function under long lasting therapy with phenprocoumon and the influence of long lasting therapy with phenprocoumon in patients suffering from aortic valve sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* 60 patients with new onset of anticoagulation therapy with phenprocoumon for the expectant duration of at least one year
* BMI 19-27 kg/qm
* Mental ability and capacity to understand and follow the instructions of the investigator
* Written informed consent

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria or with:

  * renal failure grade IV or V
  * acute cardial or pulmonary decompensation
  * women of childbearing age, pregnant or breastfeeding women
  * psychiatric diseases
  * life expectancy < 1 year
  * acute lifethreatening situations
  * participation in other studies
  * persons in dependency from the sponsor or working with the sponsor

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with required therapy with either ASS or phenprocoumon
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2008-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Progression of coronary and valvular calcification confirmed by computed tomography | 18 months

SECONDARY OUTCOMES:
Measurement of inhibitors of calcification and biomarkers for inflammation (blood samples), evaluation of the haemodynamic progress as well as dyastolic dysfunction (echocardiography) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Brandenburg, Prof., Principal Investigator — RWTH Aachen University Departement of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonology and Vascular Medicine, Aachen, North Rhine-Westphalia, Germany